CLINICAL TRIAL: NCT05532267
Title: A Randomized, Single Oral Dose, Two-way Crossover, Open-label, Laboratory Blind, Bioequivalence Study Comparing Ciprofloxacin From Two Different Drug Products After Oral Administration to Healthy Adult Subjects Under Fasting Conditions
Brief Title: Bioequivalence Study of Ciprofloxacin in Healthy Adult Subjects Under Fasting Condition
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Future University in Egypt (Other)
Responsible Party: Principal Investigator, Hala Masoud, FRC Technical Director & CEO, Future University in Egypt
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: CIP-B-20-030
Record Dates: First submitted 2022-09-04; First posted 2022-09-08 (Actual); Last update posted 2022-09-08 (Actual); Status verified 2022-09

CONDITIONS: Healthy Subjects
Keywords: Bioequivalence; Randomized; Crossover; Ciprofloxacin
MeSH Terms: interventions — Ciprofloxacin

STUDY DESIGN:
Intervention Model Description: A randomized, single-dose, two-way crossover, open-label, laboratory blind, bioequivalence study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test Product (T) (Experimental): subjects were administered a single film-coated tablet of 750 mg Ciprofloxacin with approximately 240 ml water after an overnight fast of 10 hours
  Interventions: Drug: Ciprofloxacin 750 mg
- Reference Product (R) (Active Comparator): subjects were administered a single film-coated tablet of 750 mg Ciprofloxacin with approximately 240 ml water after an overnight fast of 10 hours
  Interventions: Drug: Ciproxin 750 mg

INTERVENTIONS:
Drug: Ciprofloxacin 750 mg — an immediate release film-coated tablet containing 750 mg Ciprofloxacin
  Other Names: Test product (T)
  Arms: Test Product (T)
Drug: Ciproxin 750 mg — an immediate release film-coated tablet containing 750 mg Ciprofloxacin
  Other Names: Reference product (R)
  Arms: Reference Product (R)

SUMMARY:
To evaluate and compare the relative plasma bioavailability and therefore the bioequivalence of two different immediate release products each containing Ciprofloxacin 750 mg, after administering a single oral dose, to healthy adult subjects under fasting conditions.

DETAILED DESCRIPTION:
Enrolled subjects were randomized in a two-phase, two-sequence, cross-over design to receive a single dose of the test product (T) or the reference product (R) at each phase, under fasting conditions, with a wash-out period of 7 days.

Ciprofloxacin plasma concentrations were determined using a validated LC-MS-MS method, followed by Pharmacokinetics, and statistical analysis using Phoenix WinNonlin® software to determine the average bioequivalence.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent is obtained for study.
* Age 18 - 55 years,
* Body mass index between 18.5 and 30 kg/m2
* Have no clinically significant diseases captured in the medical history or evidence of clinically significant findings on physical examination.
* Vital signs without significant deviations.
* All laboratory screening results are within the normal range or clinically non-significant

Exclusion Criteria:

* History or presence of any disorder or condition that would render the subject unsuitable for the study, place the subject at undue risk or interfere with the ability of the subject to complete the study in the opinion of the investigator.
* History of any significant cardiovascular, hepatic, renal, respiratory, gastrointestinal, endocrine, immunologic, allergic, dermatologic, hematologic, neurologic, or psychiatric disease, or cancer.
* Any confirmed significant allergic reactions against any drug or multiple allergies.
* Clinically significant illness 28 days before study phase I.
* Alcohol or any solvent intake.
* Regular use of medication.
* Positive urine screening of drugs of abuse.
* Use of any systemic medications (prescription medications, OTC products, supplements, or herbal preparations) for 14 days prior to dosing and during the study.
* History or presence of significant smoking (more than one pack per day of cigarettes) or refusal to abstain from smoking for 48 hours before dosing until checkout.
* Blood donation within the past 60 days.
* Participation in another bioequivalence study within 60 days prior to the start of phase I of the study

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2020-11-04 (Actual); Primary Completion 2020-11-13 (Actual); Study Completion 2020-11-13 (Actual)

PRIMARY OUTCOMES:
Maximum blood concentration (Cmax) | Pre-dose (0) and at 0.25, 0.5, 0.75, 1, 1.25, 1.5, 1.75, 2, 2.25, 2.5, 2.75, 3, 3.5, 4, 5, 6, 8, 10, 12 and 24 hours after drug administration
  Cmax is observed as the maximum of ciprofloxacin peak concentration
the area under the curve (AUC 0-t) | Pre-dose (0) and at 0.25, 0.5, 0.75, 1, 1.25, 1.5, 1.75, 2, 2.25, 2.5, 2.75, 3, 3.5, 4, 5, 6, 8, 10, 12 and 24 hours after drug administration
  Cumulative Area Under the ciprofloxacin plasma concentration-time Curve calculated from 0 to time of last quantifiable concentration (t last) using the Trapezoidal method
the area under the curve extrapolated to infinity (AUC0-∞) | Pre-dose (0) and at 0.25, 0.5, 0.75, 1, 1.25, 1.5, 1.75, 2, 2.25, 2.5, 2.75, 3, 3.5, 4, 5, 6, 8, 10, 12 and 24 hours after drug administration
  AUC from Dosing time extrapolated to infinity, based on the last observed concentration

SECONDARY OUTCOMES:
Maximum time (Tmax) | Pre-dose (0) and at 0.25, 0.5, 0.75, 1, 1.25, 1.5, 1.75, 2, 2.25, 2.5, 2.75, 3, 3.5, 4, 5, 6, 8, 10, 12 and 24 hours after drug administration
  Time until Cmax is reached
Apparent terminal half-life (t½) | Pre-dose (0) and at 0.25, 0.5, 0.75, 1, 1.25, 1.5, 1.75, 2, 2.25, 2.5, 2.75, 3, 3.5, 4, 5, 6, 8, 10, 12 and 24 hours after drug administration
  the time required for the ciprofloxacin plasma concentration to decrease by 50% after the pseudo-equilibrium of distribution has been reached
Apparent elimination rate constant (Kel). | Pre-dose (0) and at 0.25, 0.5, 0.75, 1, 1.25, 1.5, 1.75, 2, 2.25, 2.5, 2.75, 3, 3.5, 4, 5, 6, 8, 10, 12 and 24 hours after drug administration
  First-order rate constant associated with the terminal (log-linear) portion of the curve

CONTACTS AND LOCATIONS:
Overall Officials: Hala Masoud, PhD, Principal Investigator — Future Research Center (FRC)
Locations (1):
- Future Research Center (FRC), Cairo, New Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this study, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol
Time Frame: Beginning 9 months following article publication and no end date
Access Criteria: Researchers who provide a methodologically sound proposal. Proposals should be directed to <hala.fut.masoud@gmail.com> To gain access.